CLINICAL TRIAL: NCT00463398
Title: Quality Control in Surgical Diagnosis and Treatment of Endometriosis.
Brief Title: Fertility Surgery, Prospective Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Christel Meuleman, MD, University Hospital, Gasthuisberg, Leuven, Belgium
Other Study IDs: ML2818 - 20/02/2006 b
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Endometriosis
Keywords: Endometriosis; Fertility Surgery; Quality of Life; Pain; Sexual Function; Health economics; Recurrence; Pregnancy
MeSH Terms: conditions — Endometriosis; Pain; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endometriosis is confirmed by histologic examination of excised lesions
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients operated at the LUFc: All patients operated at the Leuven University Fertility Centre (LUFc) between september 2006 and August 2008.

SUMMARY:
From September 2006 a prospective cohort study is conducted among all patients operated at the Leuven University Fertility Centre to evaluate clinical and economical outcome after CO2 laser laparoscopic fertility surgery.

DETAILED DESCRIPTION:
The main outcome measurements are postoperative complications, pain, quality of life, sexual satisfaction, economic life circumstances, cumulative pregnancy rate and cumulative recurrence rate of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients
* operated at the Leuven University Fertility Centre of the Department of Obstetrics and Gynaecology of the University Hospitals Leuven, Leuven,Belgium,
* from September 2006 to August 2008.

Exclusion Criteria:

* patients of other than the Dutch language

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients operated at the Leuven University Fertility Centre (LUFc) between september 2006 and August 2008.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
complication rate, quality of life, pain, sexual activity, economic life circumstances, pregnancy rate, reintervention rate, recurrence rate | 1 month preop, 6 - 12 - 18 and 24 months postop

CONTACTS AND LOCATIONS:
Overall Officials: Christel LC Meuleman, MD, Principal Investigator — University Hospital Gasthuisberg, Catholic University, Leuven, Belgium; Thomas D'Hooghe, MD, PhD, Study Director — University Hospital Gasthuisberg, Catholic University, Leuven, Belgium
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Van den Broeck U, Meuleman C, Tomassetti C, D'Hoore A, Wolthuis A, Van Cleynenbreugel B, Vergote I, Enzlin P, D'Hooghe T. Effect of laparoscopic surgery for moderate and severe endometriosis on depression, relationship satisfaction and sexual functioning: comparison of patients with and without bowel resection. Hum Reprod. 2013 Sep;28(9):2389-97. doi: 10.1093/humrep/det260. Epub 2013 Jun 24. PMID 23798058
- [Derived] Meuleman C, Tomassetti C, Wolthuis A, Van Cleynenbreugel B, Laenen A, Penninckx F, Vergote I, D'Hoore A, D'Hooghe T. Clinical outcome after radical excision of moderate-severe endometriosis with or without bowel resection and reanastomosis: a prospective cohort study. Ann Surg. 2014 Mar;259(3):522-31. doi: 10.1097/SLA.0b013e31828dfc5c. PMID 23579578